CLINICAL TRIAL: NCT03619434
Title: Pilot Study of Femtolaser Assisted Keratoplasty Versus Conventional Keratoplasty
Brief Title: Femtolaser Assisted Keratoplasty Versus Conventional Keratoplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 32158
Record Dates: First submitted 2018-07-23; First posted 2018-08-07 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Keratoconus; Fuchs Dystrophy; Corneal Disease
Keywords: Femtolaser; Corneal Transplant; Keratoplasty; Corneal Graft; Laser; Trephine
MeSH Terms: conditions — Keratoconus; Fuchs' Endothelial Dystrophy; Corneal Diseases

STUDY DESIGN:
Intervention Model Description: This is a prospective cohort study where a maximum of 30 patients attending the cornea firm at the eye unit in University Hospitals Southampton who are indicated for penetrating keratoplasty as a result of corneal disease or pathology will be recruited.
  All patients will receive a complete ophthalmological examination preoperatively.
  Subjects will then be divided randomly into 2 groups of 15, should we get 30 patients;
Masking Description: No masking as the investigators are assessing differences in surgical technique
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional keratoplasty group (Control) (Active Comparator): This group will undergo conventional penetrating keratoplasty with a trephine blade.
  Interventions: Procedure: Trephine blade
- Femtolaser group (Experimental): This group will undergo femtosecond laser-assisted penetrating keratoplasty.
  Interventions: Procedure: Femtosecond Laser

INTERVENTIONS:
Procedure: Femtosecond Laser — The laser will be used to make incisions in the cornea for the graft.
  Arms: Femtolaser group
Procedure: Trephine blade — A trephine blade will be used to make incisions in the cornea for the graft
  Arms: Conventional keratoplasty group (Control)

SUMMARY:
This pilot study will compare upto 15 patients undergoing femtolaser assisted keratoplasty (using CE[Conformité Européene] approved femtolaser apparatus) with upto 15 patients undergoing conventional keratoplasty with a manual trephine. Patients will be randomly assigned to either group. All keratoplasties will be penetrating keratoplasties. The following aims of this research is detailed below:

1. Does femtosecond laser assisted keratoplasty ( FLAK ) yield faster visual recovery and better long term BCVA (Best Corrected Visual Acuity)?
2. Does FLAK offer a biomechanically stronger cornea and thereby more safety and less risk of wound dehiscence?
3. Is there any difference between FLAK and conventional keratoplasty in terms of graft failure or rejection?

Follow up in best corrected visual acuity, various refraction/astigmatism measurements, intraocular pressure, graft rejection/failure rates, pachymetry and corneal hysteresis and resistance factor will be recorded at 1 day, 1 week, 1, 3 and 6 months and 1 year and 18 months postoperatively.

This study, to the investigators' knowledge will be the first randomised controlled trial in this area, the first to provide an empirical measurement to biomechanical stability of the cornea with the femtolaser, and the first done in an NHS (National Health Service) setting.

DETAILED DESCRIPTION:
Introduction The femtosecond laser has had a profound effect on refractive surgery and, more recently, on cataract surgery and cornea transplantation. The superior precision and control offered by femtosecond laser and its potential use in cornea transplantation show promise in terms of wound stability and strength.

By doing this research project the investigators aim to answer the following questions:

1. Does femtosecond laser assisted keratoplasty ( FLAK ) yield faster visual recovery and better long term BCVA?
2. Does FLAK offer a biomechanically stronger cornea and thereby more safety and less risk of wound dehiscence?
3. Is there any difference between FLAK and conventional keratoplasty in terms of graft failure or rejection?

There have been other studies that have compared femtolaser to the manual trephine in corneal transplant keratoplasty surgery. The investigators' study, to their knowledge, will be the first randomised controlled trial in this area. The majority of interventional studies comparing the two procedures are retrospective case controls. This study, will also be the first to provide an empirical measurement to the biomechanical stability of corneas that have undergone femtolaser corneal transplant. Although theorised to be better with the femtolaser, there has yet to have been a comparative study that has utilised quantitative evidence supporting this. By measuring postoperative corneal hysteresis and corneal resistance factor using an ocular response analyser, the investigators hope to be able to do that.

Recruitment, inclusion/exclusion and method Patients attending the cornea firm at the eye unit in University Hospitals Southampton who are indicated for penetrating keratoplasty as a result of corneal disease or pathology will be recruited. The participants have no connection to the university or the researcher that is known before the research starts. The aim for this study is to have a minimum of 10 patients recruited altogether and a maximum of 30.

Inclusion criteria: • Eyes with corneal opacities owing to previous corneal pathology.

Exclusion criteria: • Eyes with concomitant ocular pathology which may affect visual acuity.

• Eyes who received previous corneal grafts. Only after the patient has given their informed consent and confirmation that they meet the criteria will they be formally included in the study.

After inclusion in the study participants will be randomised into two groups of equal numbers to either undergo femtolaser-assisted penetrating keratoplasty or to undergo conventional keratoplasty. Other than the use of instrument to make incisions for the graft on the host cornea, all other aspects of the surgery will be kept as homogenous as possible.

Patients will stay overnight or have this operation done as a day case depending on time of day the operation is done. They will then be followed up at 1 day, 1 week, 1 months, 3 months, 6 months, 12 months and 18 months in various different visual outcome measurements as well as biomechanical measures of corneal healing. The two groups will be statistically compared at each timepoint.

This study also has a further role as a pilot study to assess the feasibility of doing a study like this on a larger scale, as a randomised, controlled trial.

Consent Patients who are deemed to not have capacity will not be eligible for this study as they cannot proceed with the consent form. All staff involved in the study have appropriate training in how to judge capacity.

For those with capacity, they will read the patient information sheet first. The patient information sheet contains in layman's terms full details for potential research participants, covering issues from why the researchers are doing the study, what the researchers expect from them, the possibility of adverse effects and anonymity and confidentiality. If patients are still interested after that they will receive a consent form to be signed by them. They will be given a copy of the signed consent form to keep.

Risks, burdens and benefits Risks are explained in the patient information sheet so patients have a fully informed decision about whether to take part in the study. From the investigators point of view it is important to note these patients for this study are indicated for corneal transplant surgery - that is it is felt the benefits of a conventional surgery outweighs the normal risks of corneal transplant surgery. Femtolaser keratoplasty is not known to add any risks that is not present in conventional keratoplasty. It is CE approved for the use in creating cuts in the cornea, as the surgeons are doing for corneal transplants.

Confidentiality The nature of this study means that their details will be known to the surgeons and staff performing the surgery in data collection but these will be coded/anonymised for members of the team involved in other parts of the study, leaving the number of people who know linking details to a minimum. Any documents linking the patient's details to the code will only be the responsibility of the surgeons and their staff. The consent forms themselves will be kept inside a locked storage unit in the Southampton Eye Unit. The patients will be reassured their personal details will not be known to any of the researchers other than the surgeons and their staff that will carry out the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Eyes with corneal opacities owing to previous corneal pathology.

Exclusion Criteria:

* Eyes with concomitant ocular pathology which may affect visual acuity.
* Eyes who received previous corneal grafts.

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-12-26 (Estimated); Study Completion 2021-12-26 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | Followed up periodically for upto 18 months
  Measure of clarity of vision
Subjective refraction | Followed up periodically for upto 18 months
  A measure of refractive error
Intraocular pressure | Followed up periodically for upto 18 months
  Fluid pressure inside the eye
Corneal hysteresis | Followed up once at 3 months
  Measure of biomechanical stability of the cornea. Will be done by one machine (Ocular Response Analyser)
Corneal topography | Followed up periodically for upto 18 months
  A visual outcome measure assessing corneal curvature. Will be done using a pentacam.
Endothelial cell density | Followed up periodically for upto 18 months
  A measure of healing in the new graft
Corneal Resistance Factor | Followed up once at 3 months
  Measure of biomechanical stability of the cornea. Will be done by one machine (Ocular Response Analyser)
Keratometry | Followed up periodically for upto 18 months
  A visual outcome measure assessing corneal curvature. Will be done using a pentacam.
Pachymetry | Followed up periodically for upto 18 months
  A visual outcome measure assessing corneal thickness. Will be done using a pentacam,
Corneal irregularity index | Followed up periodically for upto 18 months
  A visual outcome measure assessing corneal curvature. Will be done using a pentacam.
Astigmatism | Followed up periodically for upto 18 months
  A visual outcome measure assessing corneal curvature. Will be done using a pentacam.

CONTACTS AND LOCATIONS:
Overall Officials: Parwez Hossain, B ChB, PhD, Principal Investigator — University of Southampton
Locations (1):
- Southampton Eye Unit, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided